CLINICAL TRIAL: NCT01206023
Title: Applications of Nanotechnology and Chemical Sensors for the Detection and Identification of Multiple Sclerosis by Respiratory Samples
Brief Title: Applications of Nanotechnology in Multiple Sclerosis by Respiratory Samples
Acronym: MS-NANOSE
Status: Completed | Type: Observational
Sponsor: Carmel Medical Center (Other)
Collaborators: Technion, Israel Institute of Technology (Other)
Responsible Party: Principal Investigator, Ariel Miller, Director of Multiple Sclerosis & Brain Research Center, Carmel Medical Center
Other Study IDs: Nano-MS-10
Record Dates: First submitted 2010-09-19; First posted 2010-09-21 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Breath; Diagnosis; Discrimination MS/healthy subj. via exhaled breath samples
MeSH Terms: conditions — Multiple Sclerosis; Disease | interventions — Electronic Nose

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Multiple Sclerosis: Multiple Sclerosis patients
  Interventions: Other: NA-NOSE artificial olfactory system
- Healthy controls: healthy individuals
  Interventions: Other: NA-NOSE artificial olfactory system

INTERVENTIONS:
Other: NA-NOSE artificial olfactory system — NA-NOSE is an artificial olfactory system that is based on nanomaterials and connected with machine learning. NA-NOSE can diagnosis diseases or disorders based on volatile biomarkers that are emitted from exhaled breath, blood, or from clinical tissue.
  Other Names: Electronic Nose

SUMMARY:
Multiple Sclerosis (MS) is a complex multi-factorial disease, with underlying both genetic and environmental factors. Different populations have different susceptibility. The disease is characterized by 2 main phenotypes: relapsing-remitting or progressive course. Clinical disability is due to distraction of the CNS myelin.

Repair processes are mainly noted after the acute attack - and recovery of function can be spontaneous. However, in severe attacks sometimes there is need for adding STEROID TREATMENT (6 days IV) for the acute attack.

For the long term prophylactics - following the increased understanding of the disease, in the last 10-15 years there are new immunotherapies available (COPAXON / TEVA; Interferon -beta). However these can attenuate the disease (reduce the number of relapses per year) but are not cure. Also, they are beneficial in only ~40 % of the Relapsing -Remitting patients.

Currently there are no biomarkers available for MS (other than oligoclonal IgG in the CSF - which help confirm diagnosis but require invasive procedure and are not correlated with disease activity nor response to therapy) and - monitoring of MS and its treatment is by MRI - which is expensive.

Dr Hossam Haick from the Technion developed an electronic nose based nanomaterials for diagnosis of diseases (e.g., cancer, kidney failure, etc.) via breath samples.The research hypothesis is that Biomarkers of CNS inflammation and/or neurodegeneration and/or CNS repair can be detected by "electronic nose".

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a complex multi-factorial disease, with underlying both genetic and environmental factors. Different populations have different susceptibility. The disease is characterized by 2 main phenotypes: relapsing-remitting or progressive course. Clinical disability is due to distraction of the CNS myelin (mainly oligodendrocytes) due to 3 processes:

1. Inflammation- immune cells with aberrant activity invade the brain and spinal cord and cause distraction of CNS myelin.
2. Primary neurodegeneration - without prominent inflammation
3. Repair - the inflammatory and neurodegenerative processes are followed by an attempt of the CNS to repair - however, this is partial and incomplete repair is often the basis of residual deficits and disability.

   * The acute MS attack- are considered to be due to an aberrant acute immune activation and inflammatory process in the CNS
   * The chronic accumulating disability - is considered to be due to the Neuro-degenerative process.

Repair processes are mainly noted after the acute attack - and recovery of function can be spontaneous. However, in severe attacks sometimes there is need for adding STEROID TREATMENT (6 days IV) for the acute attack.

For the long term prophylactics - following the increased understanding of the disease, in the last 10-15 years there are new immunotherapies available (COPAXON / TEVA; Interferon -beta). However these can attenuate the disease (reduce the number of relapses per year) but are not cure. Also, they are beneficial in only ~40 % of the Relapsing -Remitting patients.

Currently there are no biomarkers available for MS (other than oligoclonal IgG in the CSF - which help confirm diagnosis but require invasive procedure and are not correlated with disease activity nor response to therapy) and - monitoring of MS and its treatment is by MRI - which is expensive.

Dr Hossam Haick from the Technion developed an electronic nose based nanomaterials for diagnosis of diseases (e.g., cancer, kidney failure, etc.) via breath samples. Research hypothesis Biomarkers of CNS inflammation and/or neurodegeneration and/or CNS repair can be detected by "electronic nose".

Aim(s)

Identification of biomarkers of:

1. CNS inflammation and CNS-autoimmunity
2. Neurodegeneration
3. CNS repair o that may serve as markers for disease (vs controls), of disease activity (predicting aggressive disease course (predicting Relapse; predicting Malignant vs Benign MS); predicting response to therapy (Steroid , immunotherapies or neuroprotective agents).

Work plan outline:

Evaluate few groups clinically:

* MS patients at acute relapse pre - vs- after 7 and 30 days of steroids treatment.
* Relapsing MS patients vs Progressive MS patients vs Healthy controls.
* MS patients who are Good- vs Poor- Responders to immunotherapy When available, MRI will be used as a surrogate marker, together with the clinical assessment.

Evaluation of the Electronic Nose for Diagnosis of MS We will apply a four-phase approach in order to achieve the objectives of this research. In the first phase we will collect suitable breath samples from each patient and compare the patient data to age-adjusted healthy controls. In the second phase we will analyze the collected breath samples with the electronic nose setup. In the third phase we will carry out auxiliary chemical analysis, using gas-chromatography linked with mass spectrometry (GC-MS), of the breath samples under different aspects. The fourth phase will aim at the improvement of our electronic nose setup and will be conducted in parallel to the first three phases.

We will collect breath samples of a representative group of MS patients of all types and of age-matched controls. Our GC-MS chemical analysis will address: (1) the dependence of the MS breath biomarker levels on the type/stage of the MS disease; and (2) the effect of environmental factors such as age, diet, lifestyle (especially smoking and drinking habits) on the chemical composition of the breath. Based on the results of the GC-MS chemical analysis, we will improve and optimize our array of nanosensors setup so as to achieve: (1) maximum sensitivity to the MS biomarkers and their stage dependent concentration profiles; (2) minimum sensitivity to non-MS related changes of the chemical composition of the breath, and (3) minimum sensitivity to the major ingredients of the breath, such as water vapor. We will attempt to define MS sub-categories, supported by the information from the clinical/imaging reports, which might be relevant for clinical management, by more sophisticated statistical treatment of the collected data. Towards the end of this proof-of-concept study we will compare the performance of our electronic nose setup to the conventional MS diagnostic tools. The comparison will be done in terms of true positive, true negative, false positive, false negative, sensitivity and specificity.

ELIGIBILITY:
Inclusion Criteria:

MS patients:

1. Relapsing remitting (RRMS) meeting the clinical criteria of McDonald (Polman, Reingold et al. 2005) that presented in the MS clinic in Carmel hospital, Haifa Israel. Relapsing MS patients that never received, or have received in the past, or, are currently receiving, or, are about to commence immunomodulator treatment.
2. MS patients presenting in acute relapse and about to commence a treatment regimen of corticosteroids (IV-Methylprednisolone and oral prednisone)
3. Primary progressive (PPMS) meeting the clinical criteria of McDonald (Polman, Reingold et al. 2005)that presented in the MS clinic in Carmel hospital, Haifa Israel. Tissue will be collected as previously described.
4. Willing and able to give inform consent

Control subjects:

1. Age and gender match control individuals that do not have MS or any other condition that is defined as "autoimmune". These individuals will be recruited as "Healthy Population Reference" group.
2. Willing and able to give informed consent

Exclusion Criteria:

1. Patients age 18 or less, pregnant women
2. Presence of HIV, hepatitis or any other potentially severe and infectious disease. Healthy individual with up to third degree relatives with MS or any other autoimmune diseases.

Exclusion from the experiment during the study period:

1. Any new clinical information that is not consistent with inclusion criteria.
2. Technical problems in the performance of the tests.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients of the Multiple Sclerosis Clinic, Carmel Medical Center, Israel will be invited to participate.
  Healthy volunters accompanying patients to the clinic will be invited to participate as control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 71 (Actual)
Dates: Start 2010-11; Primary Completion 2011-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Successful discrimination between healthy and MS | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Miller, MD,Ph.D, Principal Investigator — Multiple Sclerosis Center Carmel Medical Center
Locations (1):
- MS Clinic, Carmel Medical Center, Haifa, Israel